CLINICAL TRIAL: NCT01231347
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo Controlled, Trial of AMG 479 or Placebo in Combination With Gemcitabine as First Line Therapy for Metastatic Adenocarcinoma of the Pancreas
Brief Title: QUILT-2.014: Gemcitabine and AMG 479 in Metastatic Adenocarcinoma of the Pancreas
Acronym: GAMMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NantCell, Inc. (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20060540; 20060540; GAMMA; QUILT-2.014 (Other: NantCell, Inc.)
Record Dates: First submitted 2010-10-14; First posted 2010-11-01 (Estimated); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-06

CONDITIONS: Adenocarcinoma of the Pancreas; Advanced Solid Tumors; Cancer; Cancer of Pancreas; Cancer of the Pancreas; Metastases; Metastatic Cancer; Metastatic Pancreatic Cancer; Pancreas Cancer; Pancreatic Cancer; Bone Metastases; Endocrine Cancer; Oncology; Oncology Patients; Solid Tumors; Advanced Malignancy
Keywords: pancreas; gemcitabine; metastatic; jaundice
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis; Endocrine Gland Neoplasms; Jaundice | interventions — ganitumab; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo + gemcitabine (Placebo Comparator): Arm 1: AMG 479-placebo IV days 1 and 15 plus gemcitabine 1000 mg/m2 IV days 1, 8, and 15 of a 28 day cycle
  Interventions: Drug: Placebo; Drug: gemcitabine
- AMG 479 12 mg/kg dose + gemcitabine (Experimental): Arm 2: AMG 479 12 mg/kg IV days 1 and 15 plus gemcitabine 1000 mg/m2 IV days 1, 8, and 15 of a 28 day cycle
  Interventions: Drug: AMG 479; Drug: gemcitabine
- AMG 479 20 mg/kg + gemcitabine (Experimental): Arm 3: AMG 479 20 mg/kg IV days 1 and 15 plus gemcitabine 1000 mg/m2 IV days 1, 8, and 15 of a 28 day cycle
  Interventions: Drug: AMG 479; Drug: gemcitabine

INTERVENTIONS:
Drug: AMG 479 — AMG 479 12 mg/kg administered intravenously on days 1 and 15 of a 28 day cycle
  Arms: AMG 479 12 mg/kg dose + gemcitabine
Drug: Placebo — Placebo administered intravenously on days 1 and 15 of a 28 day cycle
  Arms: Placebo + gemcitabine
Drug: AMG 479 — AMG 479 20mg/kg administered intravenously on days 1 and 15 of a 28 day cycle
  Arms: AMG 479 20 mg/kg + gemcitabine
Drug: gemcitabine — gemcitabine 1000mg/m2 administered intravenously on days 1, 8 and 15 of a 28 day cycle
  Other Names: Gemzar

SUMMARY:
AMG 479 is an investigational fully human monoclonal antibody that targets type 1 insulin-like growth factor receptor (IGF-1R). Signaling through IGF-1R plays an important role in the regulation of cell growth and survival. The primary purpose of the study is to determine if AMG 479 and gemcitabine improves overall survival as compared to placebo and gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Untreated metastatic adenocarcinoma of the pancreas
* Adequate hematologic, renal and liver function
* Eastern Cooperative Oncology Group (ECOG) 0 or 1

Exclusion Criteria:

* Prior chemotherapy or radiotherapy for pancreatic cancer
* Central nervous system metastases
* External biliary drain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2011-04-07 (Actual); Primary Completion 2012-12-12 (Actual); Study Completion 2012-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NantKWest Clinical Review Team, Principal Investigator — ImmunityBio, Inc.
Locations (131):
- United States (21):
  - Research Site, Fullerton, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Rancho Mirage, California
  - Research Site, Redondo Beach, California
  - Research Site, Santa Maria, California
  - Research Site, Chicago, Illinois
  - Research Site, Harvey, Illinois
  - Research Site, Quincy, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Durham, North Carolina
  - Research Site, Bend, Oregon
  - Research Site, Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, Paris, Texas
  - Research Site, Abingdon, Virginia
  - Research Site, Spokane Valley, Washington
- Australia (6):
  - Research Site, Kogarah, New South Wales
  - Research Site, South Brisbane, Queensland
  - Research Site, Kurralta Park, South Australia
  - Research Site, Woodville South, South Australia
  - Research Site, Bentleigh East, Victoria
  - Research Site, Parkville, Victoria
- Austria (4):
  - Research Site, Innsbruck
  - Research Site, Salzburg
  - Research Site, Steyr
  - Research Site, Vienna
- Belgium (6):
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Libramont
- Brazil (2):
  - Research Site, Salvador, Estado de Bahia
  - Research Site, Porto Alegre, Rio Grande do Sul
- Bulgaria (2):
  - Research Site, Sofia
  - Research Site, Varna
- Canada (5):
  - Research Site, Vancouver, British Columbia
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
- Czechia (4):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Herlev
  - Research Site, Odense
- Finland (3):
  - Research Site, Lahti
  - Research Site, Tampere
  - Research Site, Turku
- France (3):
  - Research Site, Brest
  - Research Site, Clermont-Ferrand
  - Research Site, Pessac
- Germany (7):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Halle
  - Research Site, Mainz
  - Research Site, Mannheim
  - Research Site, Marburg
  - Research Site, Villingen-Schwenningen
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hong Kong (3):
  - Research Site, Kowloon
  - Research Site, Shatin
  - Research Site, Tuenmen
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Miskolc
- Italy (3):
  - Research Site, Genova
  - Research Site, Messina
  - Research Site, Napoli
- Japan (5):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Kashiwa, Chiba
  - Research Site, Yokohama, Kanagawa
  - Research Site, Mitaka, Tokyo
  - Research Site, Tokyo
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Eindhoven
  - Research Site, Groningen
  - Research Site, Leiden
- Poland (5):
  - Research Site, Gdansk
  - Research Site, Konin
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Warsaw
- Portugal (3):
  - Research Site, Barreiro
  - Research Site, Lisbon
  - Research Site, Porto
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Sibiu
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Kamenitz
- Slovakia (5):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Nitra
  - Research Site, Poprad
- Research Site, Ljubljana, Slovenia
- Research Site, Seoul, South Korea
- Spain (6):
  - Research Site, Santander, Cantabria
  - Research Site, Badalona, CataluÃ±a
  - Research Site, Barcelona, CataluÃ±a
  - Research Site, Elche, Valencia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Sweden (2):
  - Research Site, Eskilstuna
  - Research Site, Uppsala
- Switzerland (3):
  - Research Site, Basel
  - Research Site, Geneva
  - Research Site, Winterthur
- Research Site, Taipei City, Taipei, Taiwan
- United Kingdom (6):
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Cottingham
  - Research Site, Leicester
  - Research Site, Manchester
  - Research Site, Northampton

REFERENCES:
- [Background] Fuchs CS, Azevedo S, Okusaka T, Van Laethem JL, Lipton LR, Riess H, Szczylik C, Moore MJ, Peeters M, Bodoky G, Ikeda M, Melichar B, Nemecek R, Ohkawa S, Swieboda-Sadlej A, Tjulandin SA, Van Cutsem E, Loberg R, Haddad V, Gansert JL, Bach BA, Carrato A. A phase 3 randomized, double-blind, placebo-controlled trial of ganitumab or placebo in combination with gemcitabine as first-line therapy for metastatic adenocarcinoma of the pancreas: the GAMMA trial. Ann Oncol. 2015 May;26(5):921-927. doi: 10.1093/annonc/mdv027. Epub 2015 Jan 21. PMID 25609246
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25609246/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo + Gemcitabine | AMG 479 12 mg/kg Dose + Gemcitabine | AMG 479 20 mg/kg + Gemcitabine
Started | 322 | 318 | 160
Completed | 90 | 78 | 43
Not Completed | 232 | 240 | 117
Not completed — Full Consent withdrawn | 19 | 19 | 11
Not completed — Lost to Follow-up | 4 | 2 | 2
Not completed — Death | 202 | 210 | 101
Not completed — other event | 7 | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Gemcitabine | AMG 479 12 mg/kg Dose + Gemcitabine | AMG 479 20 mg/kg + Gemcitabine | Total
Number analyzed (Participants) | 322 | 318 | 160 | 800
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.6) | 62.1 (9.7) | 62.7 (10.1) | 62.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 159 | 75 | 368
  Male | 188 | 159 | 85 | 432
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 34 | 19 | 14 | 67
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 0 | 7
  White | 253 | 258 | 129 | 640
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 32 | 37 | 17 | 86
Region of Enrollment [Count of Participants; unit: Participants]
  Europe | 216 | 219 | 112 | 547
  United States | 26 | 31 | 13 | 70
  Canada | 4 | 3 | 1 | 8
  Australia | 13 | 7 | 4 | 24
  Japan | 30 | 34 | 16 | 80
  North Asia | 28 | 16 | 13 | 57
  South America | 5 | 8 | 1 | 14
Metastatic adenocarcinoma of the pancreas [Count of Participants; unit: Participants] | 322 | 318 | 160 | 800

OUTCOME MEASURES:

1. Primary Outcome: Determine if the Treatment of AMG 479 at 12 mg/kg and/or 20 mg/kg in Combination With Gemcitabine Improves Overall Survival as Compared With Placebo in Combination With Gemcitabine in Subjects With Metastatic Adenocarcinoma of the Pancreas
Description: The primary endpoint of the study was OS, defined as the time from randomization to death.
Time Frame: From randomization up to 20 months
Population: Full analysis set =all randomized subjects
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AMG 479 12 mg/kg Dose + Gemcitabine | AMG 479 20 mg/kg + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 318 | 160 | 322
months | 7.0 [6.2 to 8.5] | 7.1 [6.4 to 8.5] | 7.2 [6.3 to 8.2]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from screening through 30 days after the last dose of last protocol specified therapy, up to 20 months
Description: Mortality was assessed for all randomized participants (the Full Analysis Population). Adverse Events were assessed only in participants that received at least one dose of the study drug (the Safety Population).
Arm/Group | Placebo + Gemcitabine | AMG 479 12 mg/kg Dose + Gemcitabine | AMG 479 20 mg/kg + Gemcitabine
All-Cause Mortality (participants affected / at risk) | 202/322 | 210/318 | 101/160
Serious Adverse Events (participants affected / at risk) | 33/317 | 30/315 | 18/160
Other Adverse Events (participants affected / at risk) | 312/317 | 308/315 | 159/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Gemcitabine (N=317) | AMG 479 12 mg/kg Dose + Gemcitabine (N=315) | AMG 479 20 mg/kg + Gemcitabine (N=160)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 2 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 1 | 2 | 0
Cardiogenic Shock (Cardiac disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Ileus Paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 5 | 1 | 0
General Physical Health Deterioration (General disorders) | 3 | 1 | 1
Performance Status Decreased (General disorders) | 0 | 1 | 0
Sudden Death (General disorders) | 2 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 4 | 0
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 7 | 1
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3 | 4
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0
Coma Hepatic (Nervous system disorders) | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 3
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Gemcitabine (N=317) | AMG 479 12 mg/kg Dose + Gemcitabine (N=315) | AMG 479 20 mg/kg + Gemcitabine (N=160)
Nausea (Gastrointestinal disorders) | 128 | 133 | 71
Neutropenia (Blood and lymphatic system disorders) | 109 | 117 | 52
Thrombocytopenia (Blood and lymphatic system disorders) | 94 | 126 | 54
Fatigue (General disorders) | 93 | 111 | 62
Decreased Appetite (Metabolism and nutrition disorders) | 85 | 94 | 37
Vomiting (Gastrointestinal disorders) | 72 | 89 | 46
Pyrexia (General disorders) | 69 | 67 | 43
Anaemia (Blood and lymphatic system disorders) | 76 | 64 | 36
Constipation (Gastrointestinal disorders) | 62 | 82 | 29
Diarrhoea (Gastrointestinal disorders) | 58 | 84 | 27
Abdominal Pain (Gastrointestinal disorders) | 59 | 69 | 27
Hyperglycaemia (Metabolism and nutrition disorders) | 31 | 63 | 42
Oedema Peripheral (Nervous system disorders) | 58 | 49 | 25
Alanine Aminotransferase Increased (Investigations) | 45 | 61 | 24
Aspartate Aminotransferase Increased (Investigations) | 40 | 56 | 21
Asthenia (General disorders) | 45 | 47 | 18
Rash (Skin and subcutaneous tissue disorders) | 34 | 44 | 24
Leukopenia (Blood and lymphatic system disorders) | 32 | 47 | 15
Weight Decreased (Investigations) | 29 | 27 | 23
Haemoglobin Decreased (Investigations) | 22 | 38 | 9
Platelet Count Decreased (Investigations) | 17 | 31 | 21
Abdominal Pain Upper (General disorders) | 17 | 31 | 21
Back Pain (Musculoskeletal and connective tissue disorders) | 26 | 22 | 15
Blood Alkaline Phosphatase Increased (Investigations) | 19 | 31 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 22 | 12
Insomnia (Psychiatric disorders) | 25 | 20 | 10
Dysgeusia (Respiratory, thoracic and mediastinal disorders) | 13 | 23 | 13
Hyperbilirubinaemia (Blood and lymphatic system disorders) | 11 | 24 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-09-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT01231347/Prot_SAP_000.pdf